CLINICAL TRIAL: NCT07171476
Title: Enhancement of Deficient Buccal/Labial Bone Using Bone Ring Technique and Tent Pole Technique With Simultaneous Immediate Implant Placement: A Randomized Controlled Clinical Study
Brief Title: Enhancement of Deficient Labial Bone Using Bone Ring Technique and Tent Pole Technique With Immediate Implant Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 463/2022
Record Dates: First submitted 2025-08-16; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Class II Extraction Socket; Defected Buccal Bone
Keywords: immediate implant; bone ring technique; tent pole technique

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Guided bone regeneration (Active Comparator): Traditional guided bone regeneration will be done in which a 3D guided osteotomy will be done and the implant will be inserted, then covered buccally with autogenous bone graft chips and resorbable membrane before flap suturing.
  Interventions: Procedure: Guided bone regeneration
- bone ring technique (Active Comparator): Bone ring technique will be applied in which a trephine bure will be inserted through a 3D guide to prepare the site to receive the bone ring. The osteotomy will be done through the bone ring and the implant will be inserted to fix the implant in place, then covered buccally with autogenous bone graft chips and resorbable membrane before flap suturing.
  Interventions: Procedure: bone ring technique
- tent pole technique (Active Comparator): tent pole technique will be applied in which two monocortical screws will then be inserted using 3D guide, mesial and distal to the implant and extending 3 mm outside the bone, then covered buccally with autogenous bone graft chips and resorbable membrane before flap suturing.
  Interventions: Procedure: Tent pole technique

INTERVENTIONS:
Procedure: Guided bone regeneration — traditional guided bone regeneration will be done in which a flap will be raised under local anesthesia, followed by atraumatic extraction of the tooth, after which a 3D guided osteotomy will be done and the implant will be inserted, then covered buccally with autogenous bone graft chips and resorbable membrane before flap suturing
  Arms: Guided bone regeneration
Procedure: bone ring technique — bone ring technique will be applied in which the same procedure as group A will be followed till tooth extraction, after which a trephine bure will be inserted through a 3D guide to prepare the site to receive the bone ring. The osteotomy will be done through the bone ring and the implant will be inserted to fix the implant in place, then covered buccally with autogenous bone graft chips and resorbable membrane before flap suturing.
  Arms: bone ring technique
Procedure: Tent pole technique — tent pole technique will be applied in which the same procedure same as group A will be followed till implant insertion. Two monocortical screws will then be inserted using 3D guide, mesial and distal to the implant and extending 3 mm outside the bone, then covered buccally with autogenous bone graft chips and resorbable membrane before flap suturing.
  Arms: tent pole technique

SUMMARY:
Introduction: Replacing single rooted teeth with immediate implant is quit challenging in the anterior region where the buccal bone is usually deficient, moreover the bone loss increases with the extraction of tooth and the cutting of the blood supply from the periodontal ligament. With the normal bone loss around successful implant about 0.2 mm per year, its essential to start with enough buccal bone bulk to ensure long survival of the implant.

The main disadvantage of guided bone regeneration is the inability of the membrane to protect the graft from the forces exerted during suturing of the flap at the end of the procedure and the forces exerted by the patient's muscles during mastication, leading to displacement of the bone graft. Tent pole technique suggest the use of monocortical screws to support the membrane preventing displacement of the bone graft. Bone ring technique suggest surrounding the implant by ring of bone which is fixed in place by the implant itself.

Aim: The aim of the study is to evaluate the effect of Bone Ring technique, and Tent-Pole technique on buccal/Labial bone with immediate implant placement.

Methodology: Clinical study will be done in 24 cases of single rooted teeth with deficient buccal bone and require replacement with immediate implant. The 24 cases will be divided into three groups ,8 cases each. In group A, immediate implant will be placed with traditional guided bone regeneration, in which the buccal bone will be enhanced by autogenous bone chips obtained from the symphysis area and then covered by resorbable membrane. In group B, immediate implant will be placed with bone ring technique, in which autogenous bone ring obtained from the symphysis will be placed around the implant and fixed in place by the implant itself. In group C, immediate implant will be placed with tent pole technique, in which monocortical screws will be placed to support the membrane covering the autogenous bone chips obtained from the symphysis area. the implant stability will be measured immediate after implant placement and after six months from the surgery using osstel system. The buccal bone volume changes will be measured by cone beam ct.

DETAILED DESCRIPTION:
Tooth loss is still considered an epidemic condition affecting populations in different areas of the world. Immediate implant aroused as an instant solution for tooth loss with its major advantages over the conventional implant technique including preservation of bone, better soft tissue esthetic, easier placement of implant with proper position and less number of visits with less treatment time leading to less cost.

The main obstacle facing immediate implant is the insufficient buccal bone whereas the buccal bone especially in the anterior region is usually thin cortical bone with no cancellous bone support. Deprived from the blood supply supplied by the cancellous bone support, the thin buccal cancellous bone receives blood supply only from the periosteum and the periodontal ligament of the adjacent teeth which is cut during extraction leading to further decrease in blood supply and increased bone resorption. Moreover, most of the teeth which need replacing is either periodontally or apically inflamed leading to more loss of buccal bone.

Guided bone regeneration which is defined as the use of a barrier membrane to direct the growth of new bone, has been the main key to solve the insufficient buccal bone problem. However Guided bone regeneration delays the implant placement by a period of time more than 6 months which is required by the bone to build up. To decrease the time of treatment, new researches suggested applying guided bone regeneration at the same time of placing immediate implant reducing the surgical procedures to one stage procedure. Parhiz and Refoua, in 2017 placed 27 immediate implants in sockets with buccal bone defect with appling guided bone regeneration at the same procedure. The results after 6 months showed 96.3% success rate with no suppuration or thread exposure.

The main drawback of regular guided bone regeneration is the inability of the weak membrane to protect the underlaying bone graft from the forces exerted be the flap tension during the final suturing due to insufficient soft tissue or forces exerted by the patient muscles during chewing leading to bone graft displacement and failure of bone formation. (Zhenya Su et al., 2021) Tent Pole technique suggest the use of monocortical screws to support the membrane and allow enough space for the bone graft. The monocortical screws are placed extending from the bone for few millimeters required to be augmented into bone to prevent the displacement of the membrane towards the bone. In 2020, Shah et al. studied the effect tent pole technique on 10 cases of buccally defected alveolar bone ridge. The results showed that tent pole technique is an effective in augmenting vertical bone defects. (Shah et al., 2020).In 2020, Doan et al. also came to the same results concluding that tent pole technique can increase horizontal ridge dimension with minimum complications.

Bone ring technique suggest the placement of bone ring around the crestal part of the implant. A trephine bure used to prepare the recipient site just to the same size of the bone ring prepared from wither autogenous bone, allograft or xenograft. The bone ring is then placed on the prepared recipient site and the osteotomy for the implant is done through its middle hole, considering the bone ring as a guide. The implant is then placed to fix the bone ring to the site.

In 2020, Sáez et al. did a systemic review on effectiveness of the bone ring technique and simultaneous implant. 219 bone rings blocks were included in the review and the results showed a mean bone ring survival rate of 97.26% with mean bone gain of 4.94 mm In 2020, Yuan et al. compared between bone ring technique and tent-pole technique for bone augmentation of horizontally deficient alveolar ridge in the anterior maxilla. The results showed that In-situ bone ring technique evidently increased and maintained horizontal bone mass at the alveolar ridge crest compared to tent-pole technique.

3. Research Q (RQ): Can Bone Ring technique, and Tent-Pole technique enhance deficient buccal bone after immediate implant placement?

4. Research Hypothesis, Aim, Objectives & Expected Outcomes

1. Hypothesis Alternative Hypothesis theory: There is a significant difference between three materials groups Null Hypothesis theory: There is non- significant difference between the three materials groups
2. Aim The aim of the study is to evaluate the effect of Bone Ring technique, and Tent-Pole technique on buccal bone with immediate implant placement.
3. Objectives The objective of this study is to evaluate clinically and radiographically the effect of Bone Ring technique, and Tent-Pole technique on buccal/Labial bone with immediate implant placement.
4. Expected Outcomes Both Bone Ring technique, and Tent-Pole technique can enhance buccal/Labial bone with immediate implant placement.

   5. Research Design and Methods The study will be conducted after the approval of the Research Ethics Committee (REC) of the faculty of Dentistry, Suez Canal University. All patients will be selected from the outpatient clinic of the Suez Canal University hospital

I. Methods: -

1. Study setting Randomized clinical trial will be held in the outpatient clinic of the Suez Canal University hospital.
2. Sample size calculation

   The sample size for this study was calculated according to (Charan and Biswas, 2013) used the following equation:

   N =(〖(Z_α)〗^2 * 〖(S)〗^2)/〖(d)〗^2 N = Total sample size Z_α= Is Standard normal variate and its equal 1.96 at P< 0.05 SD = Standard deviation of variable d = Absolute error or precision

   Zα SD d 1.96 4.99 2

   Total sample size N =(〖(1.96)〗^2 x〖(4.99)〗^2)/〖(2)〗^2 = 23.914≈ 24 samples

   Sixteen samples will be treated within three different materials as equal (Group A and B and C) as follow:

   Groups Descriptive samples Group A Guided bone regeneration 8 Group B Bone ring technique 8 Group C Tent pole technique 8 Total samples 24
3. Patient selection

   1. Inclusion criteria (1) Patients with physical status classified as ASA class I and class II having single rooted tooth with buccal bone defect extending less than 3 mm from the alveolar bone crest which requires replacement.

   (2) There is bone extending at least 3mm beyond the root apex.

   2. Exclusion criteria
   1. Patients with physical status classified as ASA class III, class IV and class V.
   2. buccal bone defect extending more than 3 mm from the alveolar bone crest.
   3. Smoker patient.
   4. Presence of acute or chronic infection.
   5. Buccal fenestration.
4. Diagnosis and Treatment Planning

   1. Patient history: - Patient history should include information about the patient's name, age, gender, address, chief complaint and medical history.
   2. Clinical examination: - Clinical assessment of the patients will be done in a stepwise and systematic fashion including patient's general health state, and medical condition of the patient. The tooth which requires replacement will be examined to rule out presence of infection.
   3. Radiographic examination: -

   Cone beam will be done to assess:
   1. Bone density around tooth to be replaced with implant and the grey scale obtained will be converted to Hounsfield Unit (HU) by the CBCT system.
   2. The length of buccal bone defect extending from the alveolar bone crest in millimeter
   3. Whether there is a buccal fenestration or not.
   4. length and width of root to be replaced and length and width of available bone to estimate the proper implant size.
   5. Vertical dimension and horizontal dimension of the symphysis area and the thickness of cortical bone to plane for harvesting the autogenous bone in form of bone chips or bone ring according to the group.

   4. Grouping and Surgical procedure: - the 24 implant cases will be randomly divided into 3 groups, 8 implant cases each.

   Autogenous bone will be obtained from the symphysis area. A trephine bure will be used to obtain bone ring, while auto chip maker will be used to obtain bone chips.

   In group A, traditional guided bone regeneration will be done in which a flap will be raised under local anesthesia, followed by atraumatic extraction of the tooth, after which a 3D guided osteotomy will be done and the implant will be inserted, then covered buccally with autogenous bone graft chips and resorbable membrane before flap suturing.

   In group B, bone ring technique will be applied in which the same procedure as group A will be followed till tooth extraction, after which a trephine bure will be inserted through a 3D guide to prepare the site to receive the bone ring. The osteotomy will be done through the bone ring and the implant will be inserted to fix the implant in place, then covered buccally with autogenous bone graft chips and resorbable membrane before flap suturing.

   In group C, tent pole technique will be applied in which the same procedure same as group A will be followed till implant insertion. Two monocortical screws will then be inserted using 3D guide, mesial and distal to the implant and extending 3 mm outside the bone, then covered buccally with autogenous bone graft chips and resorbable membrane before flap suturing.

   5. Postoperative Follow up: -
   1. Initial stability will be measured immediately after the implant placement and final stability will be measured 6 months after the surgery using Implant Stability Quotient (ISQ) scale to compare changes in stability.
   2. Initial quadrant CBCT will be taken immediately after the implant placement and final quadrant CBCT will be taken after 6 months from the surgery to assess the changes in bone density and in bone volume vertically and horizontally.

   6. Statistical plan

   Statistical analysis. All data will be calculated, tabulated and statistically analyzed using suitable statistical tests as follow.

   A normality test (Kolmogorov-Smirnov) will be done to check normal distribution of the samples.

   Statistical analysis will be performed using the computer program SPSS software for windows version 25.0 (Statistical Package for Social Science, Armonk, NY: IBM Corp) at significant levels < 0.05 (P- Value < 0.05).

   A) Descriptive data:

   Descriptive statistics will be calculated in the form of Mean ± Standard deviation (SD), range (Max- Min).

   B) ANOVA - test or Kruskal-Wallis test (According to the types of data) One -way ANOVA (Analysis of variance) will be used to compare between the three groups under study. Tukey's or other post hoc test will be performed for the evaluation of statistical significances among the groups. P value < 0.05 is considered be statistically significant.

   C) T- test or Mann-Whitney test (According to the types of data) Independent Student's T-test or Mann-Whitney will be performed for comparison of the mean differences between the two materials at the same method at P value < 0.05.

   7. Ethics consideration: The present research will be waived from the approval of the Research Ethics Committee (REC) of the Faculty of Dentistry, Suez Canal University since it will be conducted on 24 patients. Ethical considerations regarding patient well-being and confidentiality will be undertaken by the researcher and an informed written consent will be signed by the patients before commencing the study explaining all clinical examinations, procedures and follow up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with physical status classified as ASA class I and class II having single rooted tooth with buccal bone defect extending less than 3 mm from the alveolar bone crest which requires replacement.
* There is bone extending at least 3mm beyond the root apex.

Exclusion Criteria:

* Patients with physical status classified as ASA class III, class IV or class V.
* Buccal bone defect extending more than 5 mm from the alveolar bone crest.
* Smoker patient.
* Presence of acute or chronic infection.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Implant Stability | Initial stability will be measured immediately after implant insertion before placement of cover screw and final stability will be measured after 6 months from the surgery
  stability of the implant will be measured by using a smartpeg which will be placed over the implant and the stability of the implant will be measured using Osstel ISQ system* in Implant Stability Quotient (ISQ) value in both buccolingual and mesodistal direction with the average between the two reading being recorded.
Bone density | To compare the changes in bone density in each group, the bone density around each implant was measured in two main CBCTs, which are the immediate post-operative CBCT and the final CBC taken 6 months postoperatively.
  The same section will be fixed on the immediate post-operative CBCT and the final CBCT by taking the implant as a reference. the reference lines in both the immediate post-operative the final CBCTs will be placed in the middle of the implant at both cross-section view and panoramic view fixing the same section.
  The idea of using virtual implant is to fix the area measured whereas the area drawn manually can't be fixed in both CBCTs. The virtual implant will be chosen with the same dimension and design of the used implant, placed over the real implant in both the immediate post-operative and the final CBCTs taken 6 months postoperatively. The virtual implant placed over the real implant will then be adjusted in both axial and cross-sectional views. Using the OnDemand3D CBCT analyzing system the density of 2mm thickness of bone around the implant will be measured and converted to Housefield unit.
Buccal bone height | A) Initial change The buccal bone height in preoperative CBCT will be compared to that in the immediate postoperative CBCT B) Final change The buccal bone height in preoperative CBCT will be compared to that in 6 months postoperative CBCT
  The same cut will be fixed in a cross-sectional view with zero thickness in three CBCTs representing preoperative, immediate postoperative and 6 months postoperative. The height of the buccal bone will be measured from the buccal bone crest to a fixed anatomical structure in the three CBCTs. These fixed anatomical structures include floor of the nasal cavity and maxillary sinus in the upper jaw and inferior alveolar nerve and lower border of the mandible in the lower jaw.
Buccal bone width | A) Initial change The buccal bone width in preoperative CBCT will be compared to that in the immediate postoperative CBCT B) Final change The buccal bone width in preoperative CBCT will be compared to that in 6 months postoperative CBCT
  The maximum thickness of buccal bone in the coronal third of implant will be measured in cross sectional views with zero thickness in the three CBCTs representing preoperative, immediate postoperative and 6 months postoperative.
Full ridge width | A) Initial change The maximum ridge thickness in preoperative CBCT will be compared to that in the immediate postoperative CBCT B) Final change The maximum ridge thickness in preoperative CBCT will be compared to that in 6 months postoperative CBCT
  The maximum full ridge thickness in the coronal third of implant will be measured in fixed cross-sectional views with zero thickness in the three CBCTs representing preoperative, immediate postoperative and 6 months postoperative.

CONTACTS AND LOCATIONS:
Locations (1):
- Suez Canal University, Ismailia, Ismailia Governorate, Egypt